CLINICAL TRIAL: NCT00000900
Title: The Impact of Intercurrent Illness on HIV Viral Load
Brief Title: The Effects of Illnesses on HIV Levels in the Body
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG 891
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-04

CONDITIONS: HIV Infections
Keywords: AIDS-Related Opportunistic Infections; HIV-1; Antiviral Agents; CD4 Lymphocyte Count; Polymerase Chain Reaction; RNA, Viral; Fever; Viral Load
MeSH Terms: conditions — HIV Infections; AIDS-Related Opportunistic Infections; Fever

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Other

SUMMARY:
To describe the magnitude and duration of changes in HIV-1 RNA levels during and after an acute febrile illness. To identify factors associated with increases, i.e., type of illness ultimately diagnosed (bacterial, viral, fungal), CD4 cell count, and antiretroviral treatment regimen. To describe changes in phenotypic markers of immune activation/dysregulation of CD4 and CD8 lymphocyte subsets and their relationship to intercurrent illness. To describe changes in plasma cytokines and soluble activation markers and their relationship to plasma HIV-1 viremia during and after the onset of intercurrent illness. To characterize the viral biologic phenotype and the viral drug susceptibility genotype before, during, and after the onset of an acute febrile illness. To characterize the expression of HIV-1 co-receptors before, during, and after the onset of an acute febrile illness Repeated episodes of intercurrent infections have been postulated to be an important stimulus for progression of HIV infection. The study of intercurrent illness in patients with initially undetectable viral load removes viral load as a possible cause for virologic and immunologic changes and allows for a more direct association of the intercurrent illness with changes in viral load, viral HIV-1 phenotypes, viral HIV-1 genotypes, and T cell phenotypes. Studying intercurrent illness and viral load provides an opportunity to characterize the potentially dynamic changes not only in viral load but also in phenotypic markers of T cell activation, plasma cytokine levels, phenotypic and genotypic changes in circulating virus, and HIV-1 tropisms.

DETAILED DESCRIPTION:
Repeated episodes of intercurrent infections have been postulated to be an important stimulus for progression of HIV infection. The study of intercurrent illness in patients with initially undetectable viral load removes viral load as a possible cause for virologic and immunologic changes and allows for a more direct association of the intercurrent illness with changes in viral load, viral HIV-1 phenotypes, viral HIV-1 genotypes, and T cell phenotypes. Studying intercurrent illness and viral load provides an opportunity to characterize the potentially dynamic changes not only in viral load but also in phenotypic markers of T cell activation, plasma cytokine levels, phenotypic and genotypic changes in circulating virus, and HIV-1 tropisms.

This is a study to determine whether patients exhibit a temporary burst of viral replication or other changes in response to intercurrent febrile illness. Although there is no study treatment, patients on this study must be co-enrolled in at least 1 other ACTG antiretroviral treatment study. Plasma HIV-1 RNA and other variables are measured at the time of presentation, on Day 3, and at Weeks 1, 2, 4, 8, 16, and 24.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV-1 infection documented by any licensed ELISA test kit and confirmed by either Western blot, HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA or a second antibody test by a method other than ELISA at any time prior to study entry.
* Undetectable plasma HIV-1 RNA (by Roche Amplicor Assay) within 8 weeks prior to study entry.
* Documented temperature above 101degrees F during at least 1 of the 2 days prior to the day of screening and present on the day of screening, or documented temperature above 101 F on the day of the screening but no fever on 1 of the 2 days prior to screening.

[AS PER AMENDMENT 7/7/98:

* Documented temperature above 101degrees F on the day of the screening.]
* Co-enrollment in at least 1 other ACTG antiretroviral treatment study (NOTE:
* Co-enrollment is approved and encouraged with the following ACTG studies:
* 343, 347, 359, 368, 370, and 372). [AS PER AMENDMENT 7/7/98: Must be enrolled in either an ACTG antiretroviral therapy study or a pharmaceutical company-sponsored antiretroviral therapy study prior to entry. Co-enrolled in a non-ACTG pharmaceutical company-based study must have a baseline viral isolate accessible for use in this study.]
* Written informed consent of a parent or guardian if under 18 years of age.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Interruption of current antiretroviral therapy due to the onset of acute intercurrent illness.

Concurrent Medication:

Excluded:

* Patients receiving IL-2.

Patients with the following prior conditions are excluded:

* Change in antiretroviral therapy combination within 8 weeks prior to study entry.

Required:

* Concurrent enrollment in an ACTG antiretroviral therapy study [or, AS PER AMENDMENT 7/7/98, in a non-ACTG pharmaceutical company-sponsored antiretroviral treatment study].
* Stable antiretroviral and/or nucleoside analog therapy for 8 weeks prior to study entry.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26

CONTACTS AND LOCATIONS:
Overall Officials: Sha B, Study Chair; Currier J, Study Chair
Locations (14):
- United States (14):
  - Univ of Alabama at Birmingham, Birmingham, Alabama
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Howard Univ, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - Univ of Nebraska Med Ctr, Omaha, Nebraska
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Julio Arroyo, West Columbia, South Carolina